CLINICAL TRIAL: NCT02276612
Title: A Phase 2/3, Open-Label Study to Evaluate the Safety and Efficacy of E/C/F/TAF in HIV-1 Infected Virologically Suppressed Adolescents
Brief Title: Efficacy and Safety of Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide in HIV-1 Infected Adolescents
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-292-1515; 2014-002673-11 (EudraCT Number)
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-01

CONDITIONS: HIV
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E/C/F/TAF (Experimental): Treatment-experienced participants will receive open-label E/C/F/TAF for up to 48 weeks.
  After completion of 48 weeks of treatment, all eligible participants will be given the option to participate in an open-label extension phase to receive E/C/F/TAF until a) the participant turns 18 years old and E/C/F/TAF is commercially available for use in adults in the country the participant is enrolled, or b) E/C/F/TAF becomes commercially available for use in the participant's current age group in the country the participant is enrolled, or c) E/C/F/TAF becomes accessible to participants through an access program, or d) Gilead Sciences elects to terminate development of E/C/F/TAF in the applicable country.
  Interventions: Drug: E/C/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg fixed-dose combination (FDC) tablet administered orally once daily with food
  Other Names: Genvoya®

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) in HIV-infected virologically suppressed adolescents 12 to < 18 years of age.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently on a stable antiretroviral regimen for ≥ 6 consecutive months
* Weight ≥ 35 kg (77 lbs.)
* Plasma HIV-1 RNA levels < 50 copies/mL for ≥ 6 months
* CD4+ cell count > 100 cells/μL
* No resistance to elvitegravir (EVG), emtricitabine (FTC), lamivudine (3TC) or tenofovir (TFV)
* Hepatic transaminases (AST and ALT) ≤ 5 x upper limit of normal (ULN)
* No evidence of current hepatitis B virus (HBV) infection
* No evidence of current hepatitis C virus (HCV) infection

Note: participants from Gilead Study GS-US-162-0112 were allowed to roll over into this Study GS-US-292-1515 even if they were 18 years or older at the time of screening.

Key Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to Screening
* Evidence of active pulmonary or extra-pulmonary tuberculosis disease within 3 months of screening
* Pregnant or lactating subjects

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (4):
  - Tampa, Florida
  - Detroit, Michigan
  - New York, New York
  - Memphis, Tennessee
- South Africa (3):
  - Cape Town
  - Johannesburg
  - Soweto

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in South Africa and the United States. The first participant was screened on 03 December 2014. The last study visit occurred on 23 October 2017.
Pre-assignment Details: 68 participants were screened.
Groups:
- E/C/F/TAF (12 - 17 Years of Age): Participants 12 - 17 years of age received elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) fixed-dose combination (FDC) tablet once daily with food for 48 weeks.
  Following completion of 48 weeks of treatment, eligible participants 12 - 17 years of age received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food during the open-label extension phase.
- E/C/F/TAF (≥ 18 Years of Age): Participants 18 years of age or older received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks.
  Following completion of 48 weeks of treatment, eligible participants ≥ 18 years of age received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food during the open-label extension phase.
  Note: Participants from Gilead Study GS-US-162-0112 were allowed to roll over into this Study GS-US-292-1515 even if they were 18 years or older at the time of screening.
Period: Overall Study
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Started | 50 | 10
Completed | 46 | 10
Not Completed | 4 | 0
Not completed — Death | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF (12 - 17 Years of Age): E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks in participants 12 - 17 years of age
- E/C/F/TAF (≥ 18 Years of Age): E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks in participants 18 years of age or older
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age) | Total
Number analyzed (Participants) | 50 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (1.6) | 19 (1.2) | 16 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 3 | 35
  Male | 18 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 49 | 10 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 49 | 9 | 58
  White | 1 | 0 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 0 | 8
  South Africa | 42 | 10 | 52
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 49 | 9 | 58
  ≥ 50 copies/mL | 1 | 1 | 2
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 753 (222.5) | 776 (179.9) | 757 (214.8)
CD4 Percentage [Mean (Standard Deviation); unit: percentage] | 34.3 (6.72) | 35.9 (6.53) | 34.6 (6.66)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Serious Adverse Events
Description: The percentage of participants experiencing any treatment-emergent serious adverse event was summarized.
Time Frame: Up to Week 48
Population: Safety Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
percentage of participants | 4.0 | 0

2. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: The percentage of participants experiencing any treatment-emergent adverse event was summarized.
Time Frame: Up to Week 48
Population: Safety Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
percentage of participants | 92.0 | 100.0

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level < 50 Copies/mL at Week 24 (FDA-defined Snapshot Analysis)
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: Full Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
percentage of participants | 96.0 [86.3 to 99.5] | 100.0 [69.2 to 100.0]

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Level < 50 Copies/mL at Week 48 (FDA-defined Snapshot Analysis)
Description: The percentage of participants achieving HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Full Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
percentage of participants | 90.0 [78.2 to 96.7] | 100.0 [69.2 to 100.0]

5. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
cells/µL | -72 (189.8) | -85 (245.9)

6. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 48 | 10
cells/µL | -43 (201.1) | -41 (143.0)

7. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 50 | 10
percentage | -0.6 (5.46) | -0.6 (5.46)

8. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with on-treatment data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
Number analyzed (Participants) | 48 | 10
percentage | -0.1 (3.95) | -1.1 (7.29)

ADVERSE EVENTS:
Time Frame: Up to 128 weeks plus 30 days
Description: Safety Analysis Set: participants who were enrolled in the study and received at least 1 dose of study drug.
Groups:
- E/C/F/TAF (12 - 17 Years of Age): E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks in participants 12 - 17 years of age.
  Following completion of 48 weeks of treatment, eligible participants 12 - 17 years of age received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food during the open-label extension phase.
- E/C/F/TAF (≥ 18 Years of Age): E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food for 48 weeks in participants 18 years of age or older.
  Following completion of 48 weeks of treatment, eligible participants ≥ 18 years of age received E/C/F/TAF (150/150/200/10 mg) FDC tablet once daily with food during the open-label extension phase.
Arm/Group | E/C/F/TAF (12 - 17 Years of Age) | E/C/F/TAF (≥ 18 Years of Age)
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/10
Other Adverse Events (participants affected / at risk) | 42/50 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (12 - 17 Years of Age) (N=50) | E/C/F/TAF (≥ 18 Years of Age) (N=10)
Vomiting (Gastrointestinal disorders) | 1 | 0
Electrocution (General disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF (12 - 17 Years of Age) (N=50) | E/C/F/TAF (≥ 18 Years of Age) (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 8 | 1
Axillary pain (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Pain (General disorders) | 0 | 1
Acarodermatitis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Oral herpes (Infections and infestations) | 1 | 2
Otitis media (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 3 | 1
Sinusitis bacterial (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Urinary tract infection (Infections and infestations) | 4 | 0
Viral upper respiratory tract infection (Infections and infestations) | 7 | 0
Thermal burn (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Bone density decreased (Investigations) | 2 | 1
Vitamin D decreased (Investigations) | 7 | 0
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 6 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years